CLINICAL TRIAL: NCT00343681
Title: Immunogenicity and Safety of the Inactivated, Split-Virion Influenza Vaccine, Northern Hemisphere 2006-2007 Formulation (Intramuscular Route)
Brief Title: A Study of the Immunogenicity and Safety of the 2006-2007 Influenza Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GRT63
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Influenza; Orthomyxoviridae Infections
Keywords: Influenza; Orthomyxoviridae Infections; Orthomyxoviruses; Split-virion influenza vaccine
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Inactivated influenza vaccine (split virion)

INTERVENTIONS:
Biological: Inactivated influenza vaccine (split virion) — 0.5 mL, Intramuscular

SUMMARY:
This study is designed to generate clinical data as outlined in the Note for Guidance on harmonization requirements for influenza vaccine marketing authorization by the European Medicines Agency.

The objectives of the trial are:

* To evaluate the compliance, in terms of immunogenicity, of the inactivated, split-virion influenza vaccine Northern Hemisphere 2006-2007 formulation with the requirements of the European Medicines Agency
* To describe the safety of the inactivated, split-virion influenza vaccine, Northern Hemisphere 2006-2007 formulation.

ELIGIBILITY:
Inclusion Criteria:

* Aged at least 18 years on the day of inclusion
* Informed consent form signed
* Able to attend all scheduled visits and to comply with all trial procedures
* For a woman, inability to bear a child or negative urine pregnancy test at Visit 1
* For a woman of child-bearing potential: use of an effective method of contraception or abstinence for at least four weeks prior to vaccination and at least three weeks after vaccination.

Exclusion Criteria:

* Febrile illness (oral temperature >=37.5°C) on the day of vaccination
* Breast-feeding
* Participation in another clinical trial in the four weeks preceding the trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding six months, or long-term systemic corticosteroids therapy
* Systemic hypersensitivity to egg proteins, chick proteins, or to any of the vaccine components, or history of a life-threatening reaction to the trial vaccine or a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion
* Current abuse of alcohol or drug addiction that may interfere with the subject's ability to comply with trial procedures
* Blood or blood-derived products received in the past three months
* Any vaccination in the four weeks preceding the trial vaccination
* Vaccination planned in the three weeks following the trial vaccination
* Vaccination against influenza in the previous six months
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the immunogenicity of inactivated influenza vaccine (split virion) | 21 Days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc
Locations (2):
- Allschwil, Switzerland
- Edinburgh, United Kingdom

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com